CLINICAL TRIAL: NCT03126539
Title: Effect of Topical Sulforaphane on Skin Fragility Seen in Skin Aging and With Ultraviolet Exposure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: For administrative reasons, we started a new study
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00105668
Record Dates: First submitted 2017-04-07; First posted 2017-04-24 (Actual); Results first posted 2020-02-25 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Aging
Keywords: aging; ultraviolet exposure; skin fragility; sulforaphane
MeSH Terms: interventions — sulforaphane; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Sulforaphane will be applied topically to both sites for up to 7 consecutive nights. Biopsies will be obtained prior to, and immediately after this intervention, on standard photoprotected and photoexposed sites.
  Interventions: Drug: Sulforaphane; Procedure: 4 mm skin punch biopsy
- Group B (Experimental): Two photoprotected sites will be identified. Sulforaphane will be applied topically to a single selected site for up to 7 consecutive nights. Both site will be exposed to UV. Biopsies of both sites will be obtained prior to, and 24 hours after UV exposure.
  Interventions: Drug: Sulforaphane; Radiation: Narrow-band Ultraviolet B exposure; Procedure: 4 mm skin punch biopsy

INTERVENTIONS:
Drug: Sulforaphane — Isothiocyanate sulforaphane (SF), derived from broccoli sprouts, has been known to induce an antioxidant response through the Keap1-Nrf2-antioxidant response element pathway.
  Other Names: Broccoli sprout extract; isothiocyanate sulforaphane
Radiation: Narrow-band Ultraviolet B exposure — The investigators will use a Lumera ultraviolet B (UVB) light phototherapy device which allows for targeted delivery of controlled doses of UVB radiation (emission spectrum 290-320 nm).
  Other Names: UVB, UV
  Arms: Group B
Procedure: 4 mm skin punch biopsy — All areas will be biopsied using standard punch biopsy tools and following standard clinical protocols, including cleansing the skin with an alcohol wipe and injecting local anesthesia with lidocaine and epinephrine. No more than four total skin biopsies will be obtained from a volunteer over the course of the study. After removal of the tissue sample, one or two sutures are placed to close the circular opening. Sutures are removed and a scar is formed, but typically heals well without complications and blends well with the surrounding skin.
  Other Names: biopsy

SUMMARY:
This study aims to compare the expression of keratins before and after application of sulforaphane (SF) to determine whether this agent alters skin fragility seen in both intrinsic and extrinsic skin aging and UV light exposure.

DETAILED DESCRIPTION:
The primary purpose of the study is to compare the expression of keratins before and after application of sulforaphane (SF) and determine whether these findings alter skin fragility seen in both intrinsic and extrinsic skin aging as well as in ultraviolet (UV) light exposure.

This investigation will be done in collaboration with researchers from the Department of Biochemistry and Molecular Biology and Bloomberg School of Public Health at Johns Hopkins University. The study population recruited by Johns Hopkins Department of Dermatology will include up to 50 individuals over the age of 18 with healthy skin. Each study participant will have four on-site study visits and will be asked to contribute photographs, undergo non invasive elasticity measurements, use topical sulforaphane for 7 days and contribute up to four biopsy specimens for laboratory study. The investigators will also evaluate any differences in keratins' expression in skin exposed to acute UV light, separately and after pretreatment with sulforaphane.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be over the age of 18 years old with healthy skin;
2. Must be healthy enough to undergo skin biopsy, UV light irradiation, and other study procedures in the opinion of the investigator;
3. Must be willing to comply with the requirements of the protocol;
4. Must have the ability to understand and communicate with the investigator;
5. Participant must provide informed consent.

Exclusion Criteria:

1. Subjects who are unable to provide informed consent;
2. Subject with significant medical history or current skin diseases that the investigator feels is not safe for study participation;
3. Subjects who have been treated with systemic retinoids or steroids within the past month prior to entry to the study;
4. Subjects who have been treated with topical steroids, retinoids or other topical drugs used within 2 weeks prior to entry to the study;
5. Recently treated or current skin diseases that would affect clinical evaluation and biopsy;
6. Subjects with a known allergy to broccoli.
7. Presence or suspicion of bleeding disorder or diathesis which would complicate biopsy.
8. Subjects with a history of excessive scar or keloid formation in the past 10 years.
9. Pregnant or nursing subjects (self-reported).
10. Subjects with known allergy to anesthetics used.
11. Patients with history of investigational drug use in the 30 days prior to entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chien, Principal Investigator — Johns Hopkins University
Locations (1):
- Cutaneous Translational Research Program, Department of Dermatology, Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Skin spot
Groups:
- Group A: No UV Exposure - Sulforaphane: One photoexposed site will be identified. 500nmol Sulforaphane in jojoba oil will be applied topically to site every night for up to 7 consecutive nights. Biopsy will be obtained after this intervention on standard photoexposed site.
  4 mm skin punch biopsy: All areas will be biopsied using standard punch biopsy tools and following standard clinical protocols, including cleansing the skin with an alcohol wipe and injecting local anesthesia with lidocaine and epinephrine. No more than five total skin biopsies will be obtained from a volunteer over the course of the study. After removal of the tissue sample, one or two sutures are placed to close the circular opening. Sutures are removed and a scar is formed, but typically heals well without complications and blends well with the surrounding skin.
- Group A: No UV Exposure - Placebo: One photoexposed site will be identified. Jojoba oil will be applied topically to site every night for up to 7 consecutive nights. Biopsy will be obtained after this intervention on standard photoexposed site.
  4 mm skin punch biopsy: All areas will be biopsied using standard punch biopsy tools and following standard clinical protocols, including cleansing the skin with an alcohol wipe and injecting local anesthesia with lidocaine and epinephrine. No more than five total skin biopsies will be obtained from a volunteer over the course of the study. After removal of the tissue sample, one or two sutures are placed to close the circular opening. Sutures are removed and a scar is formed, but typically heals well without complications and blends well with the surrounding skin.
- Group A: No UV Exposure - No Treatment Control: One photoprotected site and two photoexposed sites will be identified. No treatment will be administered at this site. A 4mm punch biopsy will be obtained from this site as a control.
  4 mm skin punch biopsy: All areas will be biopsied using standard punch biopsy tools and following standard clinical protocols, including cleansing the skin with an alcohol wipe and injecting local anesthesia with lidocaine and epinephrine. No more than five total skin biopsies will be obtained from a volunteer over the course of the study. After removal of the tissue sample, one or two sutures are placed to close the circular opening. Sutures are removed and a scar is formed, but typically heals well without complications and blends well with the surrounding skin.
- Group B With UV Exposure - Sulforaphane: One photoprotected site will be identified. 500nmol sulforaphane in jojoba oil will be applied topically to the site for up to 7 consecutive nights. Site will be exposed to UV. Biopsy of site will be obtained prior to, and 24 hours after UV exposure. Narrow-band Ultraviolet B (UVB) exposure: The investigators will use a Lumera UVB light phototherapy device which allows for targeted delivery of controlled doses of UVB radiation (emission spectrum 290-320nm). 4 mm skin punch biopsy: All areas will be biopsied using standard punch biopsy tools and following standard clinical protocols, including cleansing the skin with an alcohol wipe and injecting local anesthesia with lidocaine and epinephrine. No more than four total skin biopsies will be obtained from a volunteer over the course of the study. After removal of the tissue sample, one or two sutures are placed to close the circular opening. Sutures are removed and typically heals well without complications.
- Group B With UV Exposure - Placebo: One photoprotected sites will be identified. Jojoba Oil will be applied topically to a single selected site for up to 7 consecutive nights. Site will be exposed to UV. Biopsies of site will be obtained prior to, and 24 hours after UV exposure. Narrow-band Ultraviolet B (UVB) exposure: The investigators will use a Lumera UVB light phototherapy device which allows for targeted delivery of controlled doses of UVB radiation (emission spectrum 290-320nm). 4 mm skin punch biopsy: All areas will be biopsied using standard punch biopsy tools and following standard clinical protocols, including cleansing the skin with an alcohol wipe and injecting local anesthesia with lidocaine and epinephrine. No more than four total skin biopsies will be obtained from a volunteer over the course of the study. After removal of the tissue sample, one or two sutures are placed to close the circular opening. Sutures are removed and a scar is formed, but typically heals well without complications.
Period: Overall Study
Arm/Group | Group A: No UV Exposure - Sulforaphane | Group A: No UV Exposure - Placebo | Group A: No UV Exposure - No Treatment Control | Group B With UV Exposure - Sulforaphane | Group B With UV Exposure - Placebo
Started | 9; 9 Skin spot | 9; 9 Skin spot | 9; 27 Skin spot | 0; 0 Skin spot (Group B was not done) | 0; 0 Skin spot
Completed | 8; 8 Skin spot | 8; 8 Skin spot | 8; 24 Skin spot | 0; 0 Skin spot | 0; 0 Skin spot
Not Completed | 1; 1 Skin spot | 1; 1 Skin spot | 1; 3 Skin spot | 0; 0 Skin spot | 0; 0 Skin spot
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We did not enroll any participants in Group B.
Groups:
- Group A: No UV Exposure: Two photoprotected sites will be identified. Sulforaphane will be applied topically to both sites for up to 7 consecutive nights. Biopsies will be obtained prior to, and immediately after this intervention, on standard photoprotected and photoexposed sites.
  4 mm skin punch biopsy: All areas will be biopsied using standard punch biopsy tools and following standard clinical protocols, including cleansing the skin with an alcohol wipe and injecting local anesthesia with lidocaine and epinephrine. No more than four total skin biopsies will be obtained from a volunteer over the course of the study. After removal of the tissue sample, one or two sutures are placed to close the circular opening. Sutures are removed and a scar is formed, but typically heals well without complications and blends well with the surrounding skin.
- Group B With UV Exposure: Two photoprotected sites will be identified. Sulforaphane will be applied topically to a single selected site for up to 7 consecutive nights. Both site will be exposed to UV. Biopsies of both sites will be obtained prior to, and 24 hours after UV exposure.
  Narrow-band Ultraviolet B exposure: The investigators will use a Lumera UVB light phototherapy device which allows for targeted delivery of controlled doses of UVB radiation (emission spectrum 290-320 nm).
  4 mm skin punch biopsy: All areas will be biopsied using standard punch biopsy tools and following standard clinical protocols, including cleansing the skin with an alcohol wipe and injecting local anesthesia with lidocaine and epinephrine. No more than four total skin biopsies will be obtained from a volunteer over the course of the study. After removal of the tissue sample, one or two sutures are placed to close the circular opening. Sutures are removed and a scar is formed, but typically heals well without complications
- Total: Total of all reporting groups
Arm/Group | Group A: No UV Exposure | Group B With UV Exposure | Total
Number analyzed (Participants) | 9 | 0 | 9
Age, Continuous [Median (Full Range); unit: years] — Population: the same
  years | 57 [52 to 77] |  | 57 [52 to 77]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: the same
  Participants
    Female | 7 |  | 7
    Male | 2 |  | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 9 |  | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Clinical Change Score for Mottled Hyperpigmentation
Description: Clinical assessment of mottled hyperpigmentation pre and post Sulforaphane (SF) treatment will be done for both photoprotected and photodamaged skin treated with sulforaphane. Mottled Hyperpigmentation Score system will be applied, with scale of 0 to 4, 4= clear improvement after 1 week of SF or placebo application.
Time Frame: Clinical Change Score for Mottled Hyperpigmentation , up to 1 week
Population: We did not enroll any participant in group B. The results we got were not the comparison between no UV exposure group and UV exposure. Instead, the results were the clinical change score between the SF treated skin spots and no SF treated (placebo) skin spots of each participant.
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Skin spots
Arm/Group | Group A: No UV Exposure - Sulforaphane | Group A: No UV Exposure - Placebo | Group A: No UV Exposure - No Treatment Control | Group B With UV Exposure - Sulforaphane | Group B With UV Exposure - Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 0 | 0
Number analyzed (Skin spots) | 8 | 8 | 24 | 0 | 0
score on a scale | 2.8 (0.4) | .94 (.2) | 0 (0) |  |

2. Secondary Outcome: Gene Expression Changes as Assessed by Quantitative Reverse Transcription Polymerase Chain Reaction (RT-PCR)
Description: We will measure the fold-change in gene expression in human skin after acute UV light exposure, separately and in combination with application of topical sulforaphane using RT-PCR.
Time Frame: Up to 6 months
Population: Data for this outcome measure was not collected.
Arm/Group | Group A: No UV Exposure | Group B With UV Exposure
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Gene Expression Changes as Assessed by Immunohistochemistry (IHC)
Description: We will measure the fold-change in gene expression in human skin after acute UV light exposure, separately and in combination with application of topical sulforaphane using IHC.
Time Frame: Up to 6 months
Population: Data for this outcome measure was not collected.
Groups:
- Group B: Two photoprotected sites will be identified. Sulforaphane will be applied topically to a single selected site for up to 7 consecutive nights. Both site will be exposed to UV. Biopsies of both sites will be obtained prior to, and 24 hours after UV exposure.
  Sulforaphane: Isothiocyanate sulforaphane (SF), derived from broccoli sprouts, has been known to induce an antioxidant response through the Keap1-Nrf2-antioxidant response element pathway.
  Narrow-band Ultraviolet B exposure: The investigators will use a Lumera ultraviolet B (UVB) light phototherapy device which allows for targeted delivery of controlled doses of UVB radiation (emission spectrum 290-320 nm).
  4 mm skin punch biopsy: All areas will be biopsied using standard punch biopsy tools and following standard clinical protocols, including cleansing the skin with an alcohol wipe and injecting local anesthesia with lidocaine and epinephrine. No more than four total skin biopsies will be obtained from a volunteer over the c
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Four weeks
Description: We did not enroll any participants in group B.
Arm/Group | Group A: No UV Exposure | Group B With UV Exposure
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/0
Other Adverse Events (participants affected / at risk) | 0/9 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT03126539/Prot_SAP_000.pdf